CLINICAL TRIAL: NCT00943930
Title: Smoked Marijuana Discrimination and Marijuana Choice in Humans: A Laboratory Mode
Brief Title: Marijuana Drug Discrimination and Self-Administration
Acronym: DDC
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Other Study IDs: NIDA DA026761; R01DA026761-01 (NIH)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; Dextroamphetamine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Marijuana-dependent volunteers
  Interventions: Drug: THC (delta-9 tetrahydrocannabinol), d-amphetamine, oral THC

INTERVENTIONS:
Drug: THC (delta-9 tetrahydrocannabinol), d-amphetamine, oral THC — During each study session participants will be asked to smoke a cigarette. The cigarette may contain marijuana or it may contain placebo (a blank). Participants will also be asked to swallow a capsule 2-hours prior to smoking the cigarette. The capsule could contain placebo (a blank), THC (delta-9 tetrahydrocannabinol, or d-amphetamine.

SUMMARY:
This study is designed to investigate the associations among marijuana's discriminative stimulus, reinforcing, subjective (e.g. craving) and physiological effects, and to assess the relative ability of oral THC to block these effects.

DETAILED DESCRIPTION:
Volunteers will be asked to live on a research unit for up to twenty-six (26) consecutive nights and will participate in a total of 38 study sessions held on 19 weekdays. Each session will last approximately four hours and there will be two sessions per day, therefore each study day will last approximately eight hours. In addition to these study sessions, an orientation session will be conducted on the Friday prior to admission to the inpatient unit, and a lottery session will be held on the last day of the study.

During each study session participants will be asked to smoke a cigarette. The cigarette may contain marijuana or it may contain placebo (a blank). Participants will also be asked to swallow a capsule 2-hours prior to smoking the cigarette. The capsule could contain placebo (a blank), THC (delta-9 tetrahydrocannabinol, which is the active ingredient in marijuana responsible for its mood effects), or d-amphetamine. We will have participants answer questions about how the drugs make them feel and measure their vitals signs (blood pressure, heart rate, and oxygen saturation) will be measured using a non-invasive (external) vitals monitor.

ELIGIBILITY:
Inclusion Criteria:

* Female and male volunteers must be in generally good health (as indicated by results from medical history, physical exam, electrocardiogram, urine and blood samples at screening and upon arrival at the laboratory (urine samples only).
* Psychiatric examination must meet DSM-IV criteria for Cannabis Dependence.
* Individuals must be legally and mentally competent to provide written informed consent.
* Those who are unable to give their voluntary informed consent will not be accepted.

Exclusion Criteria:

* Current serious Axis I disorder (except Cannabis or Nicotine Dependence), neurologic, cardiovascular, pulmonary or systemic (e.g., renal, hepatic) disease; cognitive impairment; pregnancy (urine test), lactation (self-report), or not using (self-report) medically approved contraceptives.
* Applicants who express interest in treatment will not be accepted for study and will be provided with a treatment referral.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Marijuana dependent volunteers
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To test the ability of oral THC to alter the discriminative stimulus and reinforcing effects of smoked marijuana. | Multiple Choice Procedure Questionnaire (MCP-Q) will be administered after each drug administration sessions and participants will choose between the drug and various amounts of money.
  Three hours after each smoked marijuana dose the participant will complete the MCP-Q to make 15 independent choices between the drug dose sampled and various money amounts.

SECONDARY OUTCOMES:
Subjective effects: Self-report questionnaires regarding subjective drug effects, craving, withdrawal symptoms, and marijuana choice will be assessed. Physiological effects: Heart rate, skin temperature, and blood pressure will be monitored. | Measurements will be taken throughout a total of 40 sessions (i.e., two sessions per day) conducted over 20 weekdays. Total duration of the stay will be up to 30 days, as sessions will not be run on weekends.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States